CLINICAL TRIAL: NCT04679441
Title: : A Novel Computer-Based Functional Skills Assessment and Training Program
Brief Title: A Novel Computer-Based Functional Skills Assessment and Training Program
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: i-Function, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iFunction Phase 2
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment; Healthy Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: * Healthy individuals receive skills training only
  * MCI Participants are randomized to skills training only or skills training combined with computerized cognitive training
Who Masked: Outcomes Assessor
Masking Description: Outcomes data wil be collected in an automated manner and will be entered directly into a database
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Healthy individuals Skills training only (Active Comparator): These participants will receive CFSAT training only (n = 60). They will train for 24 hours over 12 weeks.
  Interventions: Device: The Computerized Functional Skills Assessment and Training Program
- MCI, Skills training only (Experimental): These participants will receive 24 hours of CFSAT training over 12 weeks following the same training protocol as the NC sample.
  Interventions: Device: The Computerized Functional Skills Assessment and Training Program
- MCI, Combined treatment (Experimental): Participants assigned to this condition will initially train for 3 weeks @ 60 minutes twice per week on CT (Posit Science). Participants will train 90 minutes on Double Decision and 30 minutes on Hawkeye. They can train on Hawkeye in 15- minute increments and intersperse it within the Double Decision training. They will then train CFSAT for 9 weeks at the recommended dosage. Each task will be trained twice before advancing to the next task
  Interventions: Device: The Computerized Functional Skills Assessment and Training Program; Device: Brain HQ Double Decision

INTERVENTIONS:
Device: The Computerized Functional Skills Assessment and Training Program — The CFSAT program provides training on everyday tasks critical to independent living (e.g., financial and medication management). The program currently includes six domain simulations critical to independent living: ATM Banking/Financial Management, Online Banking, Prescription Refill via Voice Menu, Kiosk Ticket Purchase, Online Shopping (and prescription refill), and Medication Management.
Device: Brain HQ Double Decision — Cognitive speed training program
  Arms: MCI, Combined treatment

SUMMARY:
People with cognitive impairments such as Mild Cognitive Impairment (MCI), often experience difficulty performing everyday routine activities. Further, normative age-related changes in cognition often lead to deficits on previously learned skills and impede new learning such as learning of new technology systems. This is of great concern, given population aging, the increasing number of older adults with cognitive impairments, and the continual deployment of new technologies in everyday contexts. The objectives of this SBIR Phase II study is to build on a previous Phase I SBIR project and refine and further evaluate a novel integrated computer-based functional skills assessment and training (CFSAT) program that provides training on everyday tasks critical to independent living (e.g., financial and medication management) with non-impaired older adults (NC) and adults with MCI.

DETAILED DESCRIPTION:
The CFSAT program provides training on everyday tasks critical to independent living (e.g., financial and medication management). The program currently includes six domain simulations critical to independent living: ATM Banking/Financial Management, Online Banking, Prescription Refill via Voice Menu, Kiosk Ticket Purchase, Online Shopping (and prescription refill), and Medication Management. The simulations are in a multi-media format and include graphic representations, voice and text. In the assessment component each of the six task domains includes subtasks that graduate in difficulty (e.g., check savings account balance, transfer money between accounts). The training component is designed to: 1) be consistent with adaptive training models of learning (tailored to the individual's skills); 2) adhere to current training guidelines for older adults, 3) identify the current levels of an individual's ability on the task with Item response theory strategies; 4) use dynamic-titration feedback from immediate task performance to adjust task difficulty to optimize training potential; and 5) provide immediate feedback and graduated instruction following errors, followed by repetition of the previously failed item. Performance metrics are captured in real time and include measures of accuracy and efficiency.

The proposed research will involve two phases and will be conducted at two locations: South Florida and New York City. Inclusion of two locations will allow us to expand the diversity of our sample and the generalizability of the findings across different regions of the U.S. Phase I will focus on validation of the 3rd alternative form of the fixed difficulty assessment tasks (form C); refinement of tasks to improve the graphical representations, enhance the difficulty level of the subtasks (based on findings from Phase 1), and ensure currency of the tasks; and usability testing of the refined tasks using a user-centered design approach. Data collection for Phase 1 will involve a sample of 24 older adults (8 non-impaired older adults aged 60+ (4 per site) and 16 with MCI aged 60+ (8 per site) (4 Spanish speaking in each group) and will take place in laboratory space at i-Function and a community location in NYC. The usability testing will occur on one day and involve approximately 2 hours. In Phase 1 the investigators will also develop browser-based version of the CFSAT program so that it can be launched from web browsers such as Google Chrome or Safari. This will greatly enhance the flexibility of the program, as the investigators will be able to launch the program from a variety of settings including the home. This is also a critical step for commercialization and direct to consumer sales.

Phase 2 will involve a multi-site trial to gather continued data on the efficacy of the CFSAT training with respect to functional gains and additional data on the usability, and acceptability of the program. The investigators will also gather data on: optimal training dosage; near and far transfer of training and environmental transfer of training (actual performance in the real world on the tasks trained by the program as tracked by the EMA protocol); the maintenance of training gains over time; the need for booster training; and adherence to home-based training protocols for those with MCI and non-impaired older adults (NC). In addition, the investigators will examine if computer-based cognitive training (CT) provides a priming effect that further enhances the benefits of the CFSAT training program for those with MCI.

ELIGIBILITY:
Inclusion Criteria MCI:

* English or Spanish speaking
* Able to read at the 6th grade level (WRAT)
* Able to read a computer screen and use a keyboard or mouse
* Has a willing and reliable informant
* Subjective memory complaints by the participant and/or collateral informant;
* Meets Jak Bondi criteria for the diagnosis of MCI.

Inclusion Criteria HC:

* Score on the MOCA ≥ 26

Exclusion Criteria:

* Sensory Limitations
* MOCA <18

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation
Enrollment: 180 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to completion on each Task of the the CFAST | Change from Baseline to end of 12 weeks of training
  Change in time to Completion time for each module
Time to completion on each Task of the the CFAST | Change from baseline to 3 months after the end of 12 weeks of training
  Change in time to Completion time for each module

SECONDARY OUTCOMES:
Performance on the Brief Assessment of Cognition App | Compared at baseline, after 12 weeks of training and 3 months after completion of training
  6-domain computerized cognitive assessments
Performance on The Virtual Reality Functional Capacity Assessment Task | Compared at baseline, after 12 weeks of training and 3 months after completion of training
  Computerized Functional Capacity Measure
EMA measurement of real world activities | For 12 weeks of training and 3 months of followup
  Participants will be surveyed as to their participation in several critical daily activities with EMA surveys

CONTACTS AND LOCATIONS:
Overall Officials: Philip Harvey, PhD, Principal Investigator — University of Miami/iFunction
Locations (2):
- United States (2):
  - Ifunction at University of Miami, Miami, Florida
  - Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
We are not planning on sharing IPD at this time as this is an SBIR

REFERENCES:
- [Result] Harvey PD, Forero DB, Ahern LB, Tibirica L, Kallestrup P, Czaja SJ. The Computerized Functional Skills Assessment and Training Program: Sensitivity to Global Cognitive Impairment, Correlations With Cognitive Abilities, and Factor Structure. Am J Geriatr Psychiatry. 2021 Apr;29(4):395-404. doi: 10.1016/j.jagp.2020.08.019. Epub 2020 Sep 7. PMID 32980252
- [Result] Harvey PD, Tibirica L, Kallestrup P, Czaja SJ. A Computerized Functional Skills Assessment and Training Program Targeting Technology Based Everyday Functional Skills. J Vis Exp. 2020 Feb 13;(156):10.3791/60330. doi: 10.3791/60330. PMID 32116309
- See also: corporate website — http://i-function.com